CLINICAL TRIAL: NCT04143464
Title: The Effectiveness of Kyphosis-specific Exercise on Reducing the Angle of Kyphosis Among Chinese Older Adults With Thoracic Hyperkyphosis - a Randomized Control Trial
Brief Title: The Effectiveness of Exercise on Reducing the Angle of Kyphosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ms Weiying Li, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: [2019] IEC (P001)
Record Dates: First submitted 2019-10-10; First posted 2019-10-29 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Kyphosis
Keywords: Thoracic Hyperkyphosis; Exercise; Older Adults
MeSH Terms: conditions — Kyphosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in this group will receive group kyphosis-specific exercise classes given by the certified physical trainer and kyphosis-specific exercise videos.
  The intervention arrangement is:
  1. Group learning and practice: a 1-hour kyphosis-specific exercise training session will be provided two times in the first week,
  2. Weekly follow-up: a 1-hour kyphosis-specific exercise will be conducted with reinforcement of learning and remedial teaching by a certified physical trainer once a week for five consecutive weeks after the group learning and practice,
  3. Self-practice: the participant will following the kyphosis-specific exercise videos doing self-practice every day for the whole intervention period lasting six weeks.
  Interventions: Behavioral: Kyphosis-specific exercise class and kyphosis-specific exercise videos
- Control group (No Intervention): No special arrangement

INTERVENTIONS:
Behavioral: Kyphosis-specific exercise class and kyphosis-specific exercise videos — The kyphosis-specific exercise is based on the protocol published by Katzman and team in 2016. It includes warm-up, back muscle strength training, spine mobility training, spine alignment training, and stretching. The class will last around 60 minutes.
  The exercise videos have the same content as the kyphosis-specific exercise class. The participants are asked to practice everyday at home following the videos.
  Arms: Intervention group

SUMMARY:
Thoracic hyperkyphosis, an exaggerated curvature between the first thoracic vertebra body (T1) and the 12th thoracic vertebra body (T12), has a high prevalence among older adults. The cross-sectional study conducted by the Principal Investigator found 72% of older adults in the Chinese community have thoracic hyperkyphosis.

Thoracic kyphosis has been found having negative effects on self-image, physical function, respiratory function, pain, balance, and gait performance. Treatment options of thoracic hyperkyphosis included surgery, peptides injection, menopausal hormone therapy, bracing, traditional Chinese medicine therapies, and exercise.

The previous studies reported that different types of exercise such as strength training, pilates, yoga, and corrective exercise were effective in reducing the thoracic hyperkyphosis. However, the previous studies either excluded older adults who have exercise habits or lack of information about participants' daily activity levels. Besides, all the group spine exercise interventions in previous studies were delivered by professional trainers or physical therapists in the form of face-to-face exercise classes.

The current RCT will be conducted to provide kyphosis-specific exercise in the form of short video and face to face exercise classes as the intervention to Chinese older adults with thoracic hyperkyphosis. The RCT can test the effects of such kyphosis-specific exercise intervention on the angle of kyphosis, physical performance, pain, and self-image among Chinese older adults with thoracic hyperkyphosis. The investigator hypotheses that older adults receive kyphosis-specific exercise intervention (video and exercise class) have reduced the angle of kyphosis. And older adults receive kyphosis-specific exercise intervention (video and exercise class) have decreased pain, better self-image, and improved overall physical performance.

DETAILED DESCRIPTION:
Thoracic hyperkyphosis, an exaggerated curvature between the first thoracic vertebra body (T1) and the 12th thoracic vertebra body (T12), has a high prevalence among older adults. The cross-sectional study conducted by the Principal Investigator found 72% of older adults in the Chinese community have thoracic hyperkyphosis.

Thoracic kyphosis has been found having negative effects on self-image, physical function, respiratory function, pain, balance, and gait performance. Treatment options of thoracic hyperkyphosis included surgery, peptides injection, menopausal hormone therapy, bracing, traditional Chinese medicine therapies, and exercise.

The previous studies reported that different types of exercise such as strength training, pilates, yoga, and corrective exercise were effective in reducing the thoracic hyperkyphosis. However, the previous studies either excluded older adults who have exercise habits or lack of information about participants' daily activity levels. Besides, all the group spine exercise interventions in previous studies were delivered by professional trainers or physical therapists in the form of face-to-face exercise classes.

The exercise protocol used by the current RCT was based on that developed by Katzmen and team. The previous studies using the same protocol reported three to five degrees decrease in the angle of kyphosis. Current RCT provides kyphosis-specific exercise in the form of short video and face to face exercise classes. The intervention of the proposed study contains two parts. One is the group kyphosis-specific exercise class given by a certified physical trainer. Another is the home practice following kyphosis-specific exercise videos. The intervention arrangement is : 1. Group learning and practice: a 1-hour kyphosis-specific exercise training session will be provided two times in the first week; 2. Weekly follow-up: a 1-hour kyphosis-specific exercise will be conducted with reinforcement of learning and remedial teaching by a certified physical trainer once a week for five consecutive weeks after the group learning and practice; 3. Self-practice: the participant will following the kyphosis-specific exercise videos doing self-practice every day for the whole intervention period lasting 6 weeks.

The group kyphosis-specific exercise class will be led by a licensed physical trainer and a trained assistant. The participant to instructor (assistant) ratio will no less than 5:1. The content of kyphosis-specific exercise videos is the same as an exercise class.

The participants are to be selected from the communities located in different regions in Wuhan by convenient sampling. Every potential participant will have a trained research assistant responsible for explaining the RCT details with the information sheet and re-assuring the respondents that data collected in the study will be kept strictly confidential, and then seeking permission for conducting the screening. The potential participants will be screened according to inclusion and exclusion criteria. The eligible participants will sign the written consent and accomplish the baseline questionnaire and assessments (T0). After that, the participant will be randomly divided into the intervention group or the control group.

A block randomization method will be used. The investigator will randomly select block sizes such as two, four, or six, to make randomization sequences for 156 participants (sample size calculation results). Then randomization sequences will be printed and placed in a sequentially numbered opaque sealed envelope. After older adult sign consent and finishing the baseline questionnaire and assessments, the researcher will open the envelope according to the numbered sequence for the grouping allocation.

The intervention group will receive a group kyphosis-specific exercise class, kyphosis-specific exercise video, and a logbook. Before every exercise class, the researcher will send them time and location as reminders. Class attendance is recorded every time. The participants are asked to record the time of home kyphosis-specific exercise practice and other daily exercises. The participants will also be encouraged to write down questions or comments in the logbook. The investigator will check the logbook and respond once a week. The Control group will receive a booklet introducing general health education material, and a logbook recording the time of daily exercises. After the end of 6 weeks of intervention, all participants will be invited to finish the postintervention assessment (T1). The data will be analyzed according to the intention to treat after T0 and T1.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese;
2. Aged 60 years and above;
3. No cognitive impairment or communication problems;
4. The angle of thoracic kyphosis > 40° measured by Manual Inclinometer;
5. Able to decrease the angle of kyphosis of 5° while standing.

Exclusion Criteria:

1. Having central or peripheral neuropathy (this may affect balance);
2. Taking drugs that affect the nervous system or affect balance and strength;
3. Having untreated severe heart and lung disease (this may affect cardiopulmonary function);
4. Having a history of spinal fracture (this may increase the risk of injury);
5. Having surgery in spinal, shoulder, and pelvis in the past year or having plan to do so in the coming six month (this may increase the risk of injury);
6. Having scoliosis ≥ 10°;
7. Having done any specific therapeutic exercise for posture in the past year or having plan to do so in the coming six month (may affect the study result).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The change of the angle of kyphosis in degrees | Baseline and after six weeks' intervention
  Measured by manual inclinometer which have previously demonstrated excellent levels of inter-rater (ICC=0.90), and intra-rater reliability (ICC=0.92), and satisfied concurrent validity (r=0.86).

SECONDARY OUTCOMES:
The time change of one leg standing in seconds (Balance) | Baseline and after six weeks' intervention
  Measured by One-leg Standing Test
The time change of up and go by seconds (Balance) | Baseline and after six weeks' intervention
  Measured by Timed Up & Go Test
The bust change in breathing by centimeters (Cardiopulmonary function) | Baseline and after six weeks' intervention
  Measured by Thoracic Expansion test
The distance change of walking by meters (Cardiopulmonary function) | Baseline and after six weeks' intervention
  the Six Minutes Walking Test
The gait performance change by gait score | Baseline and after six weeks' intervention
  Measured by the Farsi Version of Functional Gait Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Weiying Li, Mphil, Principal Investigator — PhD student, School of Nursing, the University of Hong Kong; Yong Dai, Study Director — Supervisor Nurse, Public Health Department, Liyuan Hospital of Tongji Medical College of Huazhong University of Science & Technology
Locations (2):
- Liyuan Hospital of Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei, China
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan for sharing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT04143464/Prot_SAP_000.pdf